CLINICAL TRIAL: NCT06392243
Title: Prospective, Multicenter, ranDomized Controlled, Non-Inferior Clinical Trial to Evaluate the SafeTy and effIcacy of a Novel intraCardiac Echocardiography sysTem（DISTINCT Trial）
Brief Title: IntraCardiac Echocardiography sysTem
Acronym: DISTINCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonosemi Medical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UC002
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): In the experimental group, intracardiac and large blood vessel imaging, intracardiac Doppler flow assessment and guidance of intracardiac intervention were performed by intracardiac ultrasound imaging system of Sonosemi Medical Co., Ltd.
  Interventions: Device: Intracardiac ultrasound imaging system
- Control Group (Active Comparator): The control group was treated with SOUNDSTAR 3D Diagnostic Ultrasound catheter (SNDSTR10G) and Vivid IQ, intracardiac and macrovascular imaging of the heart, assessment of intracardiac Doppler flow, and guidance for intracardiac intervention
  Interventions: Device: Intracardiac ultrasound imaging system

INTERVENTIONS:
Device: Intracardiac ultrasound imaging system — The control group was treated with SOUNDSTAR 3D Diagnostic Ultrasound catheter (SNDSTR10G) and Vivid IQ, intracardiac and macrovascular imaging of the heart, assessment of intracardiac Doppler flow, and guidance for intracardiac intervention

SUMMARY:
To evaluate the safety and effectiveness of intracardiac ultrasound imaging system in Sonosemi Medical Co., Ltd.

DETAILED DESCRIPTION:
A prospective, multicenter, randomized controlled, non-inferiority clinical trial was designed. In the experimental group, intracardiac and large blood vessel imaging, intracardiac Doppler flow assessment and guidance of intracardiac intervention were performed by intracardiac ultrasound imaging system of Sonosemi Medical Co., Ltd. The control group was treated with SOUNDSTAR 3D Diagnostic Ultrasound catheter (SNDSTR10G) and Vivid IQ, intracardiac and macrovascular imaging of the heart, assessment of intracardiac Doppler flow, and guidance for intracardiac intervention. After meeting the entry criteria, they will be randomized by an electronic randomization system, and the researchers will conduct a clinical trial based on the results of the randomization, intracardiac and large vessel imaging, intracardiac Doppler flow assessment, and guidance of intracardiac intervention were performed in both groups

ELIGIBILITY:
Inclusion Criteria:

1. patients aged ≥18 years and ≤85 years, regardless of gender,
2. patients who planned to undergo intracardiac and macrovascular imaging, intracardiac Doppler flow assessment, and intracardiac intervention,
3. subjects who could understand the purpose of the trial, were willing to cooperate with interventional treatment and follow-up, participated in the trial voluntarily and signed a written informed consent.

Exclusion Criteria:

1. known complication of sepsis, thrombosis or severe peripheral vascular disease;
2. angina class IV CCS or NYHA Class IV cardiac function,
3. severe Coagulopathy unable to perform vascular puncture,
4. known to be severely allergic to the materials used in the study;
5. pregnant or lactating women, or those who had planned to become pregnant during the trial;
6. those who were enrolled in any other drug or medical device clinical trial and had not yet left the group;
7. other conditions that the investigator judged unsuitable for enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Excellent rate of image | 0 days after the operation
  In intracardiac and large-vessel endocardial imaging of the heart, the researchers determined the ratio of"Excellent" to"Good" ultrasound image quality

CONTACTS AND LOCATIONS:
Overall Officials: He Ben, Principal Investigator — Shanghai Chest Hospital; Chu Huimin, Principal Investigator — Ningbo No. 1 Hospital; Li Haiying, Principal Investigator — The University of Hong Kong-Shenzhen Hospital; Ma Wei, Principal Investigator — Peking University First Hospital; Ning Zhongping, Principal Investigator — Zhoupu Hospital, Pudong New Area, Shanghai, China; Zhang Xiwen, Principal Investigator — Huai'an First People's Hospital
Locations (1):
- Sonosemi Medical Co., Ltd., Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No